CLINICAL TRIAL: NCT02075229
Title: A Proposal to Evaluate Revised Indications for Cochlear Implant Candidacy for the Adult CMS Population
Brief Title: Evaluation of Revised Indicatons (ERID) for Cochlear Implant Candidacy for the Adult CMS Population
Status: Completed | Type: Observational
Sponsor: American Cochlear Implant Alliance (Other)
Collaborators: University of Michigan (Other); University of Iowa (Other); Johns Hopkins University (Other); University of Miami (Other); NYU Langone Health (Other); University of North Carolina (Other); University of Southern California (Other); Vanderbilt University (Other); University of Washington (Other); Washington University School of Medicine (Other); Loyola University Chicago (Other); University of Pennsylvania (Other); University of Texas (Other); Saint Luke's Health System (Other); Massachusetts Eye and Ear Infirmary (Other); Medical College of Wisconsin (Other); Medical University of South Carolina (Other); Ohio State University (Other); Rocky Mountain Ear Center Audiology and Ear Services (Unknown)
Responsible Party: Principal Investigator, Teresa A. Zwolan, PhD, Professor and Director, University of Michigan Cochlear Implant Program, American Cochlear Implant Alliance
Other Study IDs: CAG-00107N
Record Dates: First submitted 2014-02-21; First posted 2014-03-03 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Bilateral Sensorineural Hearing Loss
Keywords: Cochlear Implant; Post-lingual onset hearing loss; Profound hearing loss; Low Frequency hearing loss; Profound sensorineural hearing loss; High frequency hearing loss; CMS-eligible patients
MeSH Terms: conditions — Hearing Loss, High-Frequency | interventions — Cochlear Implants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: 45 participants with AzBio baseline sentence scores between 41 - 50%
  Interventions: Device: Cochlear implant
- Group B: 45 participants with AzBio baseline sentence scores between 51 - 60%.
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant — A cochlear implant consists of an implantable device that electrically stimulates surviving nerve fibers within the inner ear to produce perceptions of sound in patients with significant sensorineural hearing loss.. The implanted device is controlled by an external sound processor that converts acoustic sound signals into patterns of electrical stimulation that result in sound perception for the user.

SUMMARY:
Purpose: The purpose of this study is 1) to evaluate the safety and efficacy of currently available multichannel cochlear implant systems for newly implanted adults with an indication based on open-set sentence recognition that expand criteria currently used by Center for Medicare & Medicaid Services (CMS), and 2) to assess the correlation between measures of speech recognition in candidates for cochlear implants and their utility in predicting audiologic and quality of life outcomes after implantation.

Participants: Adults (≥ 65 years of age) and CMS-eligible as a primary source of medical insurance coverage.

Procedures (methods): Evaluate objective and subjective outcomes of cochlear implantation in a patient population that does not meet current CMS candidacy criteria.

DETAILED DESCRIPTION:
Informed Consent will be obtained prior to enrollment in the study, and will include an interview to discuss study expectations, potential risks and benefits and the study evaluation schedule. The Informed Consent Form may be taken home and reviewed by the candidate and the candidate will be given the opportunity to ask questions about it and/or the study prior to signing the form. The candidate will then be given a copy of the signed Informed Consent Form.

The Informed Consent Forms will include a detailed list of procedures included in the pre-operative evaluation process. The Informed Consent document will be reviewed and signed by the relevant parties prior to any study-related evaluation taking place. Testing completed as part of normal clinical practice, such as the audiogram is acceptable prior to signing the consent form.

Information regarding each participant's hearing history will be collected and may be obtained from the participant directly or from their medical record.

The Preoperative evaluation includes:

1. Assessment of the candidate's suitability for the study
2. Establishment of baseline data if the candidate proves to be appropriate for study inclusion.

During preoperative testing, the patient will utilize hearing aids that have been verified as appropriate by the participant's managing audiologist. Clinicians will base the appropriateness of the hearing aid fitting on the recommendations of the American Academy of Audiology Task Force (2006). This includes real ear measures to verify accuracy of the hearing aid settings.

Candidacy Assessment will include

1. Air conduction thresholds for each ear with insert earphones at 125, 250, 500, 750, 1000, 1500, 2000, 3000,4000, 6000, and 8000 Hertz (Hz) Bone conduction thresholds for each ear at 125, 250, 500, 750, 1000, 1500, 2000, 4000Hz
2. AzBio Sentences Test (Quiet) - One complete recorded list at 60 dB(A) presented to the sound field with the right ear aided, left ear aided, and bilateral aided while using amplification that has been verified as appropriate by the participant's managing audiologist.

Baseline Measures Speech Perception Testing will include

1. Consonant Nucleus Consonant (CNC) Monosyllabic Word Test (Quiet) - One complete recorded list presented at 60 dB(A) in the conditions of right ear aided, left ear aided, bilateral aided
2. Telephone Testing will be performed using the ear to be implanted pre- implant. City of New York (CUNY) Sentences will be administered via live voice while the participant couples the ear to be implanted to his/her hearing aid using settings typical for phone use by that participant. If the participant is unable to use the phone, the test will still be administered with the telephone placed over the hearing aid microphone. No additional assistive listening devices (i.e. handset amplifier) or speaker phone settings will be used. Stimuli will be presented a single time only and feedback will not be provided. The examiner will use a conversational level and rate. The participant will repeat as much of the sentence as possible, guessing when necessary. Sentences will be scored for number of words repeated correctly and a percent of total words correct will be calculated.

4. Self-Assessment Questionnaires: Patients will be instructed to complete three questionnaires as they pertain to how they presently hear in everyday listening situations. These questionnaires will also be administered 6 and 12 months post-activation. :

* Health Utility Index (HUI3)
* Short Form-36 with utility transforms
* Abbreviated Profile of Hearing Aid Benefit (APHAB) Form A

Surgical Procedure: The recommended surgical procedure as outlined in the appropriate surgical manual for the device selected for implantation (provided by the device manufacturer) will be followed by the surgeon.

Postoperative Procedures will be tailored to the needs of the patient, and will vary depending on the type of cochlear implant the patient receives.

Activation should take place 2-4 weeks following surgery, or as soon as the surgeon has determined that the patient is able to participate in such an appointment and should include the following:

* Check incision site for signs of irritation or infection. Perform otoscopy. Refer patient to cochlear implant surgeon if there are concerns.
* Check adhesion of the speech processor magnet to ensure appropriateness of magnet strength. Increase or decrease magnet strength as needed.
* Perform listening check of speech processor microphone.
* Perform impedance testing (Telemetry)
* Recommended mapping parameters are provided to clinicians as defaults to begin with, but may be modified as needed based upon the recipient's response to sound.

The scheduled follow up appointments for recipients will vary depending on the recipient's response to sound, clinic schedule, and distance traveled to the clinic by the recipient. In addition to device activation, it is recommended the audiologist try to meet with patients one, three, six, and twelve months post-activation. Formal testing will be performed six and twelve months post-activation per the study protocol.

Recommended procedures to include in each mapping appointment have been provided to audiologists and include discussion of experience using the device, clarification of any questions regarding device use, listening check of speech processor microphone, impedance telemetry, psychophysical measures,loudness balancing,creation of new speech processor programs if levels have changed, and informal assessment of speech recognition.

Patients should be referred to a speech-language pathologist for formal aural rehabilitation/training if, at the three month interval he/she demonstrates no open-set speech recognition of numbers, colors, or sentences; demonstrates difficulty adjusting to the sound quality of the cochlear implant; if there is a question regarding the presence of coexisting communication difficulties related to a change in cognitive status rather than hearing impairment; or if the recipient requests additional rehabilitation and training that the audiologist is not able to provide.

Post-operative assessments will be performed at the six and twelve month test intervals and will include:

1. Audiometric Testing to include aided cochlear implant sound field warble tone thresholds at 250, 500, 1000, 2000, 3000, and 4000 Hz (if a hearing aid is used, the hearing aid will be removed and the contralateral ear will be plugged with a foam plug)
2. Speech Perception Testing will be performed with the CI alone and/or when using the CI + HA (if patient reports utilizing a hearing aid in the ipsilateral or contralateral ear at least 4 hours each day). Test will include the CNC Word Test (Quiet) - one complete list presented at 60 dB(A), and AzBio Sentences in Quiet - one complete list presented at 60 dB (A). Formal evaluation of performance using the hearing aid alone is not included in this study. Testing will include measures to evaluate performance when using the implant alone and when the patient utilizes a hearing aid plus the cochlear implant if the recipient reports that he/she utilizes a hearing aid (either in the ipsilateral or contralateral ear) a minimum of 4 hours each day. These measures include administration of CNC Words and AZ Bio Sentences in the bimodal condition of CI+HA at the 6 and 12 month post-activation intervals.
3. Self-Assessment Questionnaires described above will be re-administered six and twelve months post-activation. Patients will be instructed to complete each questionnaire as it pertains to how they presently hear in everyday listening situations (e.g. when using the CI alone or when using the CI + HA if they use a hearing aid with the CI at least 4 hours each day).
4. Telephone testing as described above but using CI alone.

Clinicians will provide participants with traditional rehabilitation, such as orientation to the device, description of strategies to improve hearing, use of assistive devices and accessories to improve performance, listening and communicating over the telephone, and counseling regarding speech recognition outcomes and expectations for performance. Audiologists will provide written materials regarding sources for independent rehabilitation and training.

RISKS AND BENEFITS The pre-specified success criteria for this protocol will be determined based on sentence recognition performance in the best aided condition. Individual levels of margin of effectiveness will be assessed based on post-operative scores on CNC Words and AZ Bio Sentences. A statistically significant improvement in pre- to postoperative performance (six to twelve months postactivation) on scores in the best aided condition will be based on the binomial distribution of Thorton and Raffin, 1978 and the binomial distribution model provided by Spahr et al., 2011.

Risks involved within this study include, but are not limited to, the risks associated with all cochlear implant surgery. It is anticipated that all study participants may permanently lose any residual hearing in the ear to be implanted. The potential benefits of cochlear implantation include improvement in the participant's ability to understand speech in quiet and in noise, with or without lip-reading, and to better detect speech and other environmental sounds.

To monitor device safety (reported through adverse events), medical and audiological observations and procedures, such as adverse device effects and unanticipated adverse device effects, are to be reported to the center's Institutional Review Board (IRB) and also to the study coordinating center. Information on all device malfunctions and adverse events will be obtained from the investigational sites and maintained by event type. The surgeon and audiologist will complete a postoperative Adverse Event Questionnaire at each postoperative test interval if any adverse events have taken place. The questions in the adverse event form elicit information regarding any surgical, medical, and device-related complications for each study participant.

Adverse device effects refer to any undesirable clinical or medical occurrence associated with use of the device or participation in the study. Adverse device effects will be reported if observed, even if they were acknowledged as risk factors in the Informed Consent Form.

Unanticipated adverse device effects refer to any event not identified above that represents a serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device if that effect, problem or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application, or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.

Investigators are to inform their respective Institutional Review Boards (IRBs) and the study coordinator immediately if an unanticipated adverse device effect is suspected (no more than 10 working days after the investigator learns of the effect). If the case is determined to be an unanticipated adverse device effect, the investigator will fill out an Unanticipated Adverse Device Effect Form. The study coordinator will report the results of an evaluation of the unanticipated adverse device effect to the FDA and all other reviewing IRBs and investigators within 10 working days after first receiving notice of the event.

ELIGIBILITY:
Inclusion Criteria:

* Sixty-five years of age or older at the time of the study and CMS-eligible as primary source of medical insurance coverage.
* Bilateral moderate to profound hearing loss in the low frequencies (up to 1000 Hz) and profound sensorineural hearing loss in the high frequencies (3000 Hz and above).
* Preoperative aided sentence score in quiet greater than or equal to 40% correct but less than or equal to 60% correct in the best aided condition on recorded AzBio sentences.
* English spoken as the primary language.

Exclusion Criteria:

* Congenital hearing loss (for the purpose of this study, onset pror to 2 years-of-age).
* Preoperative aided sentence score less than 40% or greater than 60% correct in the best aided condition on AzBio sentences in quiet
* Ossification, absence of cochlear development or any other cochlear anomaly that might prevent complete insertion of the electrode array.
* Hearing loss of neural or central origin (e.g., deafness due to lesions on the acoustic nerve or central auditory pathway).
* Active middle-ear infection.
* The audiologist and/or surgeon will review the study protocol with the patient prior to having him/her sign the consent form. If the patient indicates he/she is unwilling or unable to comply with all investigational requirements, he/she will not be enrolled in the study.
* Using best clinical judgment based on professional interaction with the patient and his/her family, the managing audiologist and surgeon will determine if there are any disabling cognitive limitations that would prevent the patient from providing reliable data for this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will evaluate the benefits of cochlear implantation in up to 90 CMS-eligible (medicare) adults from up to 10 study sites in the North America.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-02; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
AzBio sentence score at Baseline/Pre-Surgery, 6 and 12 months | up to 12 months post-cochlear implant.
  A list of recorded sentences presented to subjects prior to receiving a cochlear implant while they use hearing aids. Subjects repeat each word of the sentence that they can understand and are given a percent correct score based on the percentage of words correctly understood. The test is administered again after receiving a cochlear implant to determine if their ability to recognize words in sentences has improved.

SECONDARY OUTCOMES:
CNC Word Test at Baseline/Pre-Surgery, 6 and 12 months | Prior to receiving a cochlear implant and 6 and 12 months post- cochlear implant.
  Similar to the HINT sentences test, but instead a list of recorded one-syllable words are presented. The test is administered prior to and after receiving a cochlear implant to determine if their ability to recognize one syllable words has improved.
Health Utility Index Mark 3 (HUI3) Questionnaire at Baseline/Pre-Surgery, 6 and 12 months | Prior to receiving a cochlear implant and 6 and 12 months post- cochlear implant.
  The HUI is a family of generic health profiles and preference-based systems that measure health status and health-related quality of life.
Short Form Health Survey (SF-36) with utility transforms at Baseline/Pre-Surgery, 6 and 12 months | 6 and 12 months post- cochlear implant.
  This is a multi-purpose short-form health survey that provides an 8 scale profile of functional health and wellbeing as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index using utility transforms.
Abbreviated Profile of Hearing Aid Benefit (APHAB) | Prior to receiving a cochlear implant and 6 and 12 months post- cochlear implant.
  This is a 24 item self-assessment questionnaire scored in four subscales: Ease of Communication, Reverberation, Background Noise, and Aversiveness to Sounds.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa A Zwolan, Ph.D, Principal Investigator — University of Michigan & American Cochlear Implant Alliance
Locations (19):
- United States (19):
  - University of Southern California, Department of Otolaryngology, Head & Neck Surgery, Los Angeles, California
  - Rocky Mountain Ear Center, Englewood, Colorado
  - University of Miami, Miller School of Medicine, Miami, Florida
  - Loyola University Medical Center - Department of Otolaryngology - Head and Neck Surgery, Chicago, Illinois
  - University of Iowa, Otolaryngology-Head & Neck Surgery, Iowa City, Iowa
  - Johns Hopkins Listening Center, Baltimore, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - University of Michigan, Department of Otolaryngology, Head & Neck Surgery, Ann Arbor, Michigan
  - St. Luke's Midwest Ear Institute, Kansas City, Missouri
  - Washington University School of Medicine, Department of Otolaryngology, Head & Neck Surgery, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Department of Otolaryngology, Head & Neck Surgery, Chapel Hill, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Bill Wilkerson Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington, Virginia Merrill Bloedel Hearing Research Center, Seattle, Washington
  - Koss Cochlear Implant Program, Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zwolan TA, Kallogjeri D, Firszt JB, Buchman CA. Assessment of Cochlear Implants for Adult Medicare Beneficiaries Aged 65 Years or Older Who Meet Expanded Indications of Open-Set Sentence Recognition: A Multicenter Nonrandomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2020 Oct 1;146(10):933-941. doi: 10.1001/jamaoto.2020.2286. PMID 32857106